CLINICAL TRIAL: NCT03782103
Title: Clinical Evaluation of the Antimicrobial Effectiveness of Topically Applied ZuraPrep
Brief Title: In-vivo Efficacy of Patient Preoperative Prep, ZuraPrep (ZP)
Acronym: ZP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZX-ZP-0092 / 865-107
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2021-06

CONDITIONS: Surgical Skin Preparation
MeSH Terms: interventions — Ethanol; Chromogranins; chlorhexidine gluconate; citrate, isopropyl alcohol, methylene blue, parabens drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ZuraPrep (70% IPA) (Experimental): Isopropyl alcohol (IPA) 70%
  Interventions: Drug: ZuraPrep Clear Solution
- ChloraPrep (Active Comparator): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  Interventions: Drug: ChloraPrep
- ZuraPrep Vehicle (Placebo Comparator): Zurex Prep without IPA
  Interventions: Drug: ZuraPrep Vehicle

INTERVENTIONS:
Drug: ZuraPrep Clear Solution — Apply topically.
  Other Names: Isopropyl alcohol 70%; ZP
  Arms: ZuraPrep (70% IPA)
Drug: ChloraPrep — Apply topically.
  Other Names: CHG 2%/IPA 70%; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Arms: ChloraPrep
Drug: ZuraPrep Vehicle — Apply topically.
  Other Names: Vehicle
  Arms: ZuraPrep Vehicle

SUMMARY:
The objective of the study is to demonstrate the antimicrobial efficacy of the Zurex Preoperative Prep (ZuraPrep - clear) on skin flora of the abdomen and inguinal regions of human subjects.

DETAILED DESCRIPTION:
The primary objective of this study is to measure the antimicrobial effectiveness of a single investigational test article, ZuraPrep™ as specified by the Healthcare Antiseptics, Topical Antimicrobial Drug Products Final Rule of December 20, 2017. The treatments will be ZuraPrep™ as the investigational test article, ChloraPrep® as an active control, and ZuraPrep™ Vehicle as a negative control. For efficacy at 30 seconds post-prep, the test article should be superior to the negative control using a margin of 1.2 log10 CFU/cm2 and non-inferior to the active control using a margin of 0.5 log10 CFU/cm2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good general health
* Minimum bacterial baseline requirements on abdomen and groin
* Skin free of tattoos, dermatoses, abrasions, cuts, lesions, or other skin disorder near or on the applicable test area.

Exclusion Criteria:

* Topical or systemic antimicrobial exposure within 14 days prior to screening and treatment days, including antibiotics.
* Taking antihistamines, immunosuppressants, or oral steroids within 14 days prior to screening and treatment days, excluding contraception or post-menopausal treatment.
* Subjects with allergies to study materials including isopropyl alcohol or chlorhexidine gluconate.
* Subjects with a history of skin sensitivity, skin allergies, or skin cancer.
* Subjects who are pregnant, attempting pregnancy or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M H Bashir, MD, Principal Investigator — Microbac Laboratories, Inc.
Locations (1):
- Microbac Laboratories, Inc., Sterling, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment consists of subjects that advanced from screening to randomization and treatment. Each subject had 2 test products applied bilaterally; therefore, the numbers will not add up uniformly across arms due to the pre-determined cohort/block design. Result totals will be less than than the treated number as the per subject/area/intervention anatomical site must have an acceptable baseline count/flora.
Units Other Than Participants: Ab or groin
Groups:
- All Study Participants: ZP (Isopropyl alcohol (IPA) 70%) or CP or ZP Vehicle, applied topically to abdominal (for 30 seconds) or groin (for 2 minutes).
Period: Overall Study
Arm/Group | All Study Participants
Started | 156; 72 Ab or groin
ZP | 156; 72 Ab or groin
CP | 156; 72 Ab or groin
Vehicle | 156; 72 Ab or groin
Completed | 156; 72 Ab or groin
Not Completed | 0; 0 Ab or groin

BASELINE CHARACTERISTICS:
Population: Subjects must have the following bacteria counts to entry study, for the abdomen, the allowable baseline log10 CFU/cm2 value > 3.0; for the groin, the allowable baseline log10 CFU/cm2 value > 5.0.
Units Other Than Participants: Abdomen or groin
Groups:
- Treatment Population: Each subject could have received 2 out of 3 test products randomly assigned. Demographics were not stratified by test product due to study design. While 156 was the treated population, to be evaluable for efficacy, each subject anatomical sample site (4/per subject) would need to pass the minimum log10 CFU/cm2 baseline requirements.
Arm/Group | Treatment Population
Number analyzed (Participants) | 156
Number analyzed (Abdomen or groin) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 156
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.90 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 150
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 39
  Asian | 59
  Native Hawaiian or Other Pacific Islander | 17
  Black or African American | 0
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 156

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Reduction - Groin
Description: A 3-log10 CFU/cm^2 bacterial reduction on the inguinal region is considered a success.
Time Frame: 30 seconds post product application
Population: Treated subjects with a treatment day baseline criteria of 5.0-7.5 log10 CFU/cm^2 recoveries for each sampling site (2 groin sampling sites per subject).
Measure: Mean (Standard Deviation); unit: log 10 CFU/cm2
Units Other Than Participants: Abdomen or groin
Groups:
- Mean Log Reduction - ZP (70% IPA) - Groin: Isopropyl alcohol (IPA) 70%
  ZP: Apply topically.
- Mean Log Reduction - ChloraPrep - Groin: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  ChloraPrep: Apply topically.
- Mean Log Reduction - ZP Vehicle - Groin: ZP without IPA
  ZP Vehicle: Apply topically.
Arm/Group | Mean Log Reduction - ZP (70% IPA) - Groin | Mean Log Reduction - ChloraPrep - Groin | Mean Log Reduction - ZP Vehicle - Groin
Number analyzed (Participants) | 156 | 156 | 156
Number analyzed (Abdomen or groin) | 79 | 77 | 83
log 10 CFU/cm2 | 4.133 (0.4) | 3.642 (0.5) | 1.277 (0.6)
Statistical Analysis 1: Comparison: Mean Log Reduction - ZP (70% IPA) - Groin vs Mean Log Reduction - ChloraPrep - Groin; Groin 30 seconds post product application, Average Treatment Effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 CFU/cm^2 bacterial counts and the predictors were the treatment effect as a fixed effect and the pre-treatment log10 CFU/cm^2 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product upper bounds must be less than 0.5; Median Difference (Final Values) = -0.2845, 95% CI 2-sided [-0.6033 to 0.0334]
Statistical Analysis 2: Comparison: Mean Log Reduction - ZP (70% IPA) - Groin vs Mean Log Reduction - ZP Vehicle - Groin; Groin 30 seconds post product application, Average Treatment Effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 CFU/cm^2 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 CFU/cm^2 bacterial counts as a covariate; Test type: Superiority — Investigational product lower bounds must be greater than 1.2; Mean Difference (Final Values) = 2.8535, 95% CI 2-sided [2.5415 to 3.1655]

2. Primary Outcome: Bacterial Reduction - Abdomen
Description: A 2-log10 CFU/cm^2 bacterial reduction on the abdomen region is considered a success.
Time Frame: 30 seconds post product application
Population: Treated subjects with a treatment day baseline criteria of 3.0 - 5.5 Log10 CFU/cm^2 recoveries.
Measure: Mean (Standard Deviation); unit: Log10 CFU/cm^2
Units Other Than Participants: Abdomen or groin
Groups:
- Mean Log Reduction - ZP (70% IPA) - Abdomen: Isopropyl alcohol (IPA) 70%
  ZP: Apply topically.
- Mean Log Reduction - ChloraPrep - Abdomen: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  ChloraPrep: Apply topically.
- Mean Log Reduction - ZP Vehicle - Abdomen: ZP without IPA
  ZP Vehicle: Apply topically.
Arm/Group | Mean Log Reduction - ZP (70% IPA) - Abdomen | Mean Log Reduction - ChloraPrep - Abdomen | Mean Log Reduction - ZP Vehicle - Abdomen
Number analyzed (Participants) | 156 | 156 | 156
Number analyzed (Abdomen or groin) | 83 | 81 | 78
Log10 CFU/cm^2 | 3.036 (0.4) | 3.087 (0.4) | 1.234 (0.5)
Statistical Analysis 1: Comparison: Mean Log Reduction - ZP (70% IPA) - Abdomen vs Mean Log Reduction - ChloraPrep - Abdomen; Abdomen 30 seconds post product application, Average Treatment Effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 CFU/cm^2 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 CFU/cm^2 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product average treatment effect upper bounds cannot be more than 0.5; Mean Difference (Final Values) = 0.0577, 95% CI 2-sided [-0.1457 to 0.2611]
Statistical Analysis 2: Comparison: Mean Log Reduction - ZP (70% IPA) - Abdomen vs Mean Log Reduction - ZP Vehicle - Abdomen; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Investigational product lower bounds must be greater than 1.2; Mean Difference (Final Values) = 1.8208, 95% CI 2-sided [1.6153 to 2.0264]

3. Secondary Outcome: Bacterial Counts Not Exceeding Baseline in the Abdomen and Groin Region
Description: Bacterial counts should not exceed baseline on the abdomen or groin region
Time Frame: 6 hours post product applcation
Population: Subjects were treated and post treatment the 6 hour log10 CFU/cm2 values were evaluated for persistence. If the 6 hour value was below the baseline log10CFU/cm2 value, then the site had a persistent effect. This was calculated as a binary variable: 1 if the site had a persistent effect; 0 if not.
Measure: Number; unit: Abd or groin with persistent effect
Units Other Than Participants: Abdomen or groin
Groups:
- ZP (70% IPA): Isopropyl alcohol (IPA) 70% - 6 hr post product application
  ZP: Apply topically.
Arm/Group | ZP (70% IPA)
Number analyzed (Participants) | 156
Number analyzed (Abdomen or groin) | 72
Abd or groin with persistent effect | 72

ADVERSE EVENTS:
Time Frame: 6 hours post product application
Groups:
- Zurex Prep (70% IPA): Isopropyl alcohol (IPA) 70%
  ZuraGard Clear Solution: Apply topically.
- Zurex Prep Vehicle: Zurex Prep without IPA
  Zurex Prep Vehicle: Apply topically.
Arm/Group | Zurex Prep (70% IPA) | ChloraPrep | Zurex Prep Vehicle
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/156 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/156 | 0/156
Other Adverse Events (participants affected / at risk) | 0/156 | 0/156 | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03782103/Prot_SAP_000.pdf